CLINICAL TRIAL: NCT01292629
Title: Comparison of the HSO iSert 251 Posterior Chamber Aspheric Aphakic Intraocular Lens to Historical / Literature Controls.
Brief Title: Comparison of the Hoya Surgical Optics (HSO) iSert 251 Posterior Chamber Aspheric Aphakic Intraocular Lens to Historical / Literature Controls.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hoya Surgical Optics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-N251
Record Dates: First submitted 2011-02-04; First posted 2011-02-09 (Estimated); Results first posted 2015-03-20 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Aphakia; Cataract
Keywords: intraocular lens; IOL; cataract; Hoya; surgical; optics; ocular; visual acuity
MeSH Terms: conditions — Aphakia; Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Investigational intraocular lens (Experimental): iSert 251 intraocular lens
  Interventions: Device: iSert 251 intraocular lens

INTERVENTIONS:
Device: iSert 251 intraocular lens — aphakic intraocular lens

SUMMARY:
The purpose of this multi-center clinical trail is to determine the safety and efficacy of the iSert 251 for the correction of aphakia.

DETAILED DESCRIPTION:
This study evaluated the safety and effectiveness of the Hoya Surgical Optics iSert Model 251 IOL following primary implantation for the visual correction of aphakia in adults in whom the cataractous lens has been removed by phacoemulsification. Results from this prospective, multicenter clinical trial will be used to support a PMA supplement for the iSert® 251 IOL.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with cataract for which phacoemulsification extraction and posterior chamber IOL implantation is indicated
* Have clear intraocular media
* Have potential Best Corrected Visual Acuity of 20/40 or better
* Have preoperative Best Spectacle-Corrected visual acuity of 20/40 or worse

Exclusion Criteria:

* Have ocular pathology or abnormalities that do or are expected to reduce best corrected visual acuity in the operative eye during the study period
* Are monocular
* Have current ocular infection
* Are taking systemic steroids or other anti-metabolites
* Have previous retinal detachment in the operative eye or expect to require retinal laser treatment during the course of the study

Eligibility criteria not complete. Contact Hoya Surgical Optics, Inc. for more information.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2011-02; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kees den Besten, Study Director — Hoya Surgical Optics
Locations (5):
- United States (5):
  - Schwartz Laser Eye Center, E. Shea Blvd, Suite C101, Arizona
  - Katzen Eye Care and Laser Center, Boynton Beach, Florida
  - Center for Excellence in Eye Care, Miami, Florida
  - Eye Surgeons of Indiana, Indianapolis, Indiana
  - Eye Health Vision Centers, North Dartmouth, Massachusetts

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects who were >50 years of age, either sex, and any race were eligible for this study. Diagnosis of cataracts in one or both eyes.
Pre-assignment Details: Subject's eligibility was determined at the preoperative visit. All subject met inclusion/exclusion criteria.
Groups:
- iSert 251: iSert 251 Intraocular Lens: Implantation with the iSert® 251 Intraocular lens
Period: Overall Study
Arm/Group | iSert 251: iSert 251 Intraocular Lens
Started | 125
Completed | 125
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- iSert® 251 Intraocular Lens: Population Description: A total of 125 subjects were implanted with the iSert® IOL. Data analysis for baseline characteristics was completed on these 125 subjects.
Arm/Group | iSert® 251 Intraocular Lens
Number analyzed (Participants) | 125
Age, Customized [Number; unit: participants] — A total of 125 subjects were implanted with the iSert® IOL. Data analysis for baseline characteristics was completed on these 125 subjects.
  participants
    < 60 years of age | 7
    61 - 69 years of age | 50
    70 - 79 years of age | 53
    ≥ 80 years of age | 15
Sex/Gender, Customized [Number; unit: participants]
  Female | 77
  Male | 48

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity
Description: BEST Spectacle-Correction (ETDRS) Distance Visual Acuity
Time Frame: 4 to 6 months
Population: 125 subjects enrolled in the study, 121 were examined at the Form 4 and the remaining four (3.2%) subjects missed the Form 4 visit but were examined later. 121 subjects were evaluated for primary and secondary effectiveness and safety outcomes.
Measure: Number; unit: subjects
Groups:
- iSert 251: iSert 251 Intraocular Lens: Eligible subjects underwent phacoemulsification cataract extraction surgery and were implanted with the iSert® Intraocular Lens. Study observation was up to 271 days.
Arm/Group | iSert 251: iSert 251 Intraocular Lens
Number analyzed (Participants) | 121
subjects
  Subjects with BSCVA 20/40 or Better at Visit 3 | 121
  Subjects with BSCVA 20/40 or Better at Visit 4 | 121

2. Secondary Outcome: Complications and Adverse Events
Description: Number of Participants with Complications or Adverse Events
Time Frame: 4 to 6 months
Measure: Number; unit: participants
Groups:
- iSert 251 Aphakik IOL: iSert 251: iSert 251 intraocular lens
Arm/Group | iSert 251 Aphakik IOL
Number analyzed (Participants) | 125
participants | 0

ADVERSE EVENTS:
Time Frame: 4-6 months
Groups:
- iSert 251: iSert 251 Intraocular Lens: Subjects who underwent phacoemulsification cataract extraction surgery who were implanted with the iSert aphakic intraocular lens.
Arm/Group | iSert 251: iSert 251 Intraocular Lens
Serious Adverse Events (participants affected / at risk) | 0/125
Other Adverse Events (participants affected / at risk) | 0/125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No